CLINICAL TRIAL: NCT05483959
Title: Biphasic Positive Airway Pressure in the Management of Acute Respiratory Distress Syndrome: A Comparative Study
Brief Title: BIPAP in the Management of Acute Respiratory Distress Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Shymaa Sayed Salem, doctor, South Valley University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: BIPAP IN ARDS
Record Dates: First submitted 2022-07-25; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Mechanical Ventilation Complication
Keywords: BIPAP , ARDS

STUDY DESIGN:
Intervention Model Description: BIPAP mode of ventilation applied to 20patients , SIMV PC mode applied to the other group
Who Masked: Participant
Masking Description: Mechanically ventilated ARDS patients
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BIPAP group (Experimental): Mechanically ventilated ARDS patients on BIPAP mode of ventilation
  Interventions: Other: BIPAP mode/SIMV PC mode
- SIMV PC group (Experimental): Mechanically ventilated ARDS patients on SIMV PC mode of ventilation
  Interventions: Other: BIPAP mode/SIMV PC mode

INTERVENTIONS:
Other: BIPAP mode/SIMV PC mode — BIPAP is a mode of ventilation recently used in ARDS

SUMMARY:
Evaluation of biphasic positive airway pressure as a new mode of ventilation in management of acute respiratory failure constituted in ARDS as a category of hypoxaemic respiratory failure in comparison to conventional ventilation.

DETAILED DESCRIPTION:
Biphasic positive airway pressure (BIPAP) is a mode of mechanical ventilation that allow unrestricted spontaneous breathing independent of ventilator cycling, using an active expiratory valve. BIPAP mode is pressure-limited and time-cycled, Ventilation occurs via the time-cycled switching between two set pressure levels. In the absence of spontaneous breathing, this mode resemble conventional pressure controlled ventilation.

A proposed advantage of BIPAP compared to conventional pressure-controlled ventilation is the improved distribution of gas to dependent lung regions as the result of spontaneous breathing enabled during the inspiratory and expiratory time cycles, so prevents atelectasis and promotes alveolar recruitment resulting in an improved ventilation-perfusion matching.

ARDS is an acute diffuse, inflammatory lung injury, leading to increased pulmonary vascular permeability, increased lung weight, and loss of aerated lung tissue with hypoxemia and bilateral radiographic opacities, associated with increased venous admixture, increased physiological dead space and decreased lung compliance.

In patients with ARDS, BIPAP with spontaneous breathing contributes to improved pulmonary gas exchange, systemic blood flow and oxygen supply to the tissue. This is reflected by clinical improvement in the patient's condition, which is associated with significantly fewer days on ventilatory support, earlier extubation and a shorter stay in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* All intubated Adult ARDS patients
* ARDS is diagnosed according to berlin criteria.

Exclusion Criteria:

* Age < 18 years.
* Cardiac or respiratory arrest on admission.
* Morbid obesity with BMI > 40.
* Acute exacerbation of IPF.
* Cerebrovascular or neuro muscular disorder. 6. Diabetic ketoacidosis. 7. Hepatic or renal disease. 8.Cardiac disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-04-20 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Oxygen saturation of the participants will be measured from the arterial blood gases taken from the patient and according to the range of oxygen saturation from 90 to 98% will be compared | Baseline
  Base line oxygen saturation of BIPAP group and SIMV PC group patients will be taken from the arterial blood gases and recorded from the range of oxygen saturation from 90 to 98% and will be compared between both groups
Blood pressure in mm Hg of BIPAP group and SIMV PC group will be measured by the sphygmomanometer device | Base line
  Blood pressure in mm Hg of BIPAP group and SIMV PC group will be measured by the sphygmomanometer device and will be compared between both groups according to the normal range of systolic blood pressure from 90mmHg to 130mmHg and diastolic blood pressure from the range of 60 mmHg to 90 mmHg
Lung mechanics including the tidal volume by ml per kg ideal body weight of BIPAP and SIMV PC groups will be taken from the ventilators and recorded | 24 hours after mechanical ventilation
  Lung mechanics including the tidal volume by ml per kg ideal body weight of BIPAP and SIMV PC groups will be taken from the ventilators and compared between both groups according to the range of tidal volume from 4 to 8 ml per kg ideal body weight

SECONDARY OUTCOMES:
Duration of mechanical ventilation of BIPAP group | 6 weeks
  The duration of mechanical ventilation duration had been compared between both groups
The duration of anesthesia in days | 2 weeks
  The duration of anesthesia in days on BIPAP group willassessed between BIPAP group and SIMV PC group

CONTACTS AND LOCATIONS:
Overall Officials: Khaled H Ahmed, Professor, Study Director — Assiut University; Alaa R Mahmoud, Professor, Principal Investigator — faculty of medicine, South Valley University; Gad S Gad, Professor, Study Chair — faculty of medicine, South Valley University
Locations (1):
- Shymaa Sayed Salem, Qina, Qena Governorate, Egypt

REFERENCES:
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Hedenstierna G, Lattuada M. Gas exchange in the ventilated patient. Curr Opin Crit Care. 2002 Feb;8(1):39-44. doi: 10.1097/00075198-200202000-00007. PMID 12205405
- [Result] Hormann C, Baum M, Putensen C, Mutz NJ, Benzer H. Biphasic positive airway pressure (BIPAP)--a new mode of ventilatory support. Eur J Anaesthesiol. 1994 Jan;11(1):37-42. PMID 8143712